CLINICAL TRIAL: NCT07134426
Title: Investigating Vaped Phenanthrene Biomarkers in Former Smokers
Brief Title: Vaped Phenanthrene
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2022LS127
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Former Smoker; Non-Smoker
Keywords: Smoking; Tobacco; Vaping; Former Smoker; Non-Smoker
MeSH Terms: conditions — Smoking Cessation; Smoking; Vaping

STUDY DESIGN:
Intervention Model Description: All study participants (Former Daily Smokers and Non-smokers) will be asked to vape D10-phenanthrene to see how their lungs breakdown a class of cancer-causing chemicals known as polycyclic aromatic hydrocarbons [PAHs].
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D10-phenanthrene (Other): All study participants (Former Daily Smokers and Non-smokers) will be asked to vape D10-phenanthrene to see how their lungs breakdown a class of cancer-causing chemicals known as polycyclic aromatic hydrocarbons [PAHs].
  Interventions: Other: D10-phenanthrene

INTERVENTIONS:
Other: D10-phenanthrene — All study participants (Former Daily Smokers and Non-smokers) will be asked to vape D10-phenanthrene to see how their lungs breakdown a class of cancer-causing chemicals known as polycyclic aromatic hydrocarbons [PAHs].

SUMMARY:
Some people who used to smoke cigarettes continue to be at higher risk of developing lung cancer, even years after quitting. This study will look to see if a specific chemical, phenanthrene, is broken down in the lungs of former smokers through more harmful pathways than never-smokers. If former smokers break down chemicals that enter their lungs through more harmful pathways this might be putting them at higher risk for developing lung cancer even though they quit smoking. This information may help find better ways to prevent or treat cancer in the future.

This study is under an IND, but the drug is not being studied; instead, it is being used as a marker for drug metabolism.

ELIGIBILITY:
Inclusion Criteria:

* > 21 years of age
* In good physical & mental health
* In stable physical & mental health
* Have tried vaping
* Former daily cigarette smokers who quit 1-20 year ago
* Non-smokers who have not used tobacco or nicotine products

Exclusion Criteria:

* Has any respiratory disease (ex - asthma, COPD, etc...)
* Has/had high blood pressure
* Has/had liver disease
* Has/had cancer
* Has experience negative effects when vaped previously
* Pregnant or nursing

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Urinary Ratio of D10PheT/D9PhOH | 24 hours after vaping phenanthrene
  The ratio of D10-phenanthrene tetraol to D9-phenanthrene phenols in the urine will determine how the lung breaks down a class of cancer-causing chemicals called Polycyclic Aromatic Hydrocarbons (PAHs). The higher this ratio the more the lungs break down these chemicals through harmful pathways, which might increase cancer risk. The lower the ratio the more the lung breaks down the chemicals through safer pathways.
TNE | Baseline measure
  Total nicotine equivalents will be measured in the urine samples to confirm that study participants are not using tobacco or nicotine products.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hecht, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No